CLINICAL TRIAL: NCT05088473
Title: Diagnosic and Pronostic Values of Kappa and Lambda Free Light Chains in Central Nervous System Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Neuro01
Record Dates: First submitted 2021-07-13; First posted 2021-10-22 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Central Nervous System Diseases; Multiple Sclerosis
Keywords: multiple sclerosis; kappa free light chains; lambda free light chains
MeSH Terms: conditions — Central Nervous System Diseases; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mutliple sclerosis
  Interventions: Other: Biological collection
- CIS/RIS
  Interventions: Other: Biological collection
- Other CNS inflammatory diseases
  Interventions: Other: Biological collection
- Non inflammatory CNS diseases
  Interventions: Other: Biological collection

INTERVENTIONS:
Other: Biological collection — Collection of cerebrospinal fluid kappa and lambda free light chains and indexes

SUMMARY:
Numerous studies have shown the diagnostic interest of cerebrospinal fluid kappa free light chains and kappa index in multiple sclerosis. However, large cohort studies are lacking and little is known about the correlation between kappa and lambda indexes and multiple sclerosis evidence disease activity. Therefore, this study plan to validate the kappa and lambda free light chains and indexes as diagnostic biomarker in multiple sclerosis and to correlate the concentration of kappa and lambda free light chains with clinical and radiological activity in a large cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms evocative of CNS involvement for who serum and cerebrospinal fluid kappa free light chains and kappa index are available

Exclusion Criteria:

* Infectious CNS disease
* Tumor CNS disease
* Active CNS bleeding
* Monoclonal gammapathy
* Severe chronic renal failure (glomerular filtration rate <30 ml/mn)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with symptoms evocative of CNS disease
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Measurement of cerebrospinal fluid (CSF) and serum kappa and lambda free light chains (KFLC and LFLC) | 1 day
  1. Measurement of cerebrospinal fluid (CSF) and serum KFLC and LFLC by a turbilimetric analyzer (data in mg/L)
  2. Quantification of QKFLC and QLFLC (CSF FLC/serum FLC) in each group of patients
  3. Compare median of QKFLC and QLFLC between groups
Measurement of cerebrospinal fluid (CSF) and serum albumin | 1 day
  1. Measurement of cerebrospinal fluid (CSF) and serum albumin by the same turbilimetric analyzer (data in mg/L)
  2. Quantification of albumin quotient (AQ) (CSF albumin/serum albumin) in each group of patients
Evaluation of the diagnostic performances of KFLC and LFLC intrathecal synthesis biomarkers (K/L FLC index and K/L FLC intrathecal fraction (IF)) for multiple sclerosis | 1 day
  1. Calculation of KFLC intrathecal synthesis biomarkers:
     KFLC index = (CSF KFLC/serum KFLC) / AQ
     KFLC IF = (KFLC(loc)/CSF KFLC) x 100 with:
     KFLC(loc) = ((CSF KFLC/serum KFLC) / Qk(lim)) x serum KFLC and Qk(lim) = 3.27 x (AQ^2 + 33)^0.5 - 8.2
  2. Calculation of LFLC intrathecal synthesis biomarkers:
     LFLC index = (CSF LFLC/serum LFLC) / AQ)
     LFLC IF = (LFLC(loc)/CSF LFLC) x 100 with:
     LFLC(loc) = ((CSF LFLC/serum LFLC) / Ql(lim)) x serum LFLC and Ql(lim) = 2.1138 x AQ^0.865
  3. Determination of diagnostic performances by ROC curve analysis and best cut-off values with the Younden index to calculate sensitivity, specificity and predictive values for MS diagnosis
Comparison of diagnostic performances of K/L FLC intrathecal synthesis biomarkers to oligoclonal bands (OCB) for multiple sclerosis | 1 day
  1. Identification of OCB status for each patient
  2. Calculation of diagnostic performances of OCB (sensitivity, specificity and predictive values) for MS diagnostic
  3. Comparison of diagnostic performances (sensitivity, specificity and predictive values) of OCB and K/L FLC intrathecal synthesis biomarkers for multiple sclerosis

SECONDARY OUTCOMES:
Evaluation of clinical data that can alter KFLC and LFLC values | 1 day
  Identification of data that can be independtly associated with high or low CSF KFLC or LFLC values as potential bias in K/L FLC intrathecal synthesis biomarkers interpretation:
  * Gender
  * Age
  * Type of clinical demyelinating event (i.e. myelitis, optic neuritis...)
  * Immune modifying drug treatment ongoing during sampling
  * Underlying disease activity (measured by the presence of subacute clinical symptoms ongoing at sampling or gadolinium enhanced lesions within the last MRI status)

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Universitaire de Lille, Lille
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Assistance Publique des Hôpitaux de Paris, Paris
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier Régional et Universaitaire de Tours, Tours

IPD SHARING:
Plan to Share IPD: No